CLINICAL TRIAL: NCT07215351
Title: Impact of the Inno Cleanse Dietary Supplement on Gut Health and Associated Variables in Healthy Men and Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: INNOSUPPS (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO-FY2025-554
Record Dates: First submitted 2025-10-08; First posted 2025-10-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Constipation; Bloating
Keywords: Inno Cleanse
MeSH Terms: conditions — Constipation | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Dietary Supplement (Experimental): 15 randomly assigned individuals will receive 2 capsules daily of the experimental dietary supplement for 2 weeks with assessments prior and after intervention.
  Interventions: Dietary Supplement: Dietary supplement for digestive health
- Placebo Control (Placebo Comparator): 15 randomly assigned individuals will receive 2 capsules daily of the placebo for 2 weeks with assessments prior and after intervention.
  Interventions: Dietary Supplement: placebo capsule

INTERVENTIONS:
Dietary Supplement: Dietary supplement for digestive health — Dietary supplement contains cascara sagrada bark powder, cape aloe leaves extract, senna leaf powder, frangula bark powder fennel seed powder, bentonite clay, burdock root powder, licorice root extract, slippery elm bark powder, Capiscum annuum L. Fruit powder, milk thistle seed powder, hydroxypropyl methylcellulose, and silicon dioxide.
  Arms: Experimental Dietary Supplement
Dietary Supplement: placebo capsule — Contains hydroxypropyl methylcellulose and cellulose
  Arms: Placebo Control

SUMMARY:
The purpose of the present study is to investigate the impact of a natural dietary supplement, Inno Cleanse™, to reduce bloating in a population of otherwise healthy men and women, who claim to feel frequently bloated. Inno CleanseTM dietary supplement is manufactured in the United States under current Good Manufacturing Practices (cGMP) and is marketed by InnoSupps as a digestive health aid. It is sold in the United States on the company's website, Amazon, and in many large retail outlets. It remains a very popular product, with close to 1.4 million units sold since 2020, with a reported 66,000 units sold in the past three months.

Despite the prevalence of dietary supplements identifying as digestive aids, detoxification, and cleanses, very little research has been done to determine their effectiveness. The product appears to be well-designed, with multiple ingredients included which have scientific evidence of effectiveness. That said, and despite the overall positive reviews, there is no known clinical research to support the product's effectiveness.

Therefore, the aim of this study is to evaluate the efficacy of the Inno Cleanse product to reduce bloating and result in other positive outcomes (weight loss). This study will be run as a double-blind placebo-controlled trial, in which subjects will use the product or placebo for two weeks. It is hypothesized that treatment with the dietary supplement Inno Cleanse will result in reduced bloating, as evidenced by self-reported reductions in bloating and hunger, as well as moderate weight loss and a reduction in body circumference measures due to the reduced bloating. In addition, multiple anecdotal reports of improved skin health have been noted in those using the product. Additionally, routine blood and urine sample analysis will be performed as a secondary outcome, as a safety measure.

ELIGIBILITY:
Inclusion Criteria:

* experience regular (2 or more days per week) bloating or constipation
* able to fast a minimum of 12 hours prior to testing visit

Exclusion Criteria:

* pregnant, planning to become pregnant, or breastfeeding
* sensitivity or allergic to any components of the study product (cascara sagrada bark powder, cape aloe leaves extract, senna leaf powder, frangula bark powder fennel seed powder, bentonite clay, burdock root powder, licorice root extract, slippery elm bark powder, Capiscum annuum L. Fruit powder, milk thistle seed powder, hydroxypropyl methylcellulose, cellulose, and silicon dioxide).
* experienced a severe allergic reaction that resulted in emergency care
* diagnosed with medical disorders linked to digestive/gut health such as celiac disease, crohn's disease, gastroesophageal reflux disease, heartburn, irritable bowel syndrome, ulcerative colitis, ulcers, etcetera.
* experiencing regular diarrhea
* active infection or illness
* diabetic
* hypertensive
* cardiovascular disease
* breast, uterine, or ovarian cancer
* uterine fibroids or endometriosis
* taking medications or supplements that may alter gut health including but not limited to diuretics, laxatives, anti-diarrheal, anticholinergic agents, or antispasmodic agents.
* previous adverse experience with laxatives
* taking medications known to interact with the dietary supplement's ingredients including blood pressure medications, anticoagulants, antiplatelets, blood thinners, cholesterol-lowering medications, diuretics, water pills, estrogen based contraceptives, non-steroidal anti-inflammatory drugs, digoxin, corticosteroids, Monoamine oxidase inhibitors, insulin, medications processed in the liver, diclofenac, fluvastatin, glipizide, ibuprofen, piroxicam, phenytoin, phenobarbital, or secobarbital.
* tobacco user
* strenuous activity within 24 hours of testing visits
* caffeine within 24 hours of testing visit
* alcohol within 24 hours of testing visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Alanine transaminase | baseline
  Alanine transaminase measured as part of metabolic panel in international units per liter
Alanine transaminase | 2 weeks of assigned intervention
  Alanine transaminase measured as part of metabolic panel in international units per liter
Aspartate transferase | baseline
  Aspartate transferase measured as part of metabolic panel in international units per liter
Aspartate transferase | 2 weeks of assigned intervention
  Aspartate transferase measured as part of metabolic panel in international units per liter
Albumin | baseline
  Albumin measured as part of metabolic panel in grams per deciliter
Albumin | 2 weeks of assigned intervention
  Albumin measured as part of metabolic panel in grams per deciliter
Alkaline phosphatase | baseline
  Alkaline phosphatase measured as part of metabolic panel in international units per liter
Alkaline phosphatase | 2 weeks of assigned intervention
  Alkaline phosphatase measured as part of metabolic panel in international units per liter
Total bilirubin | baseline
  Total bilirubin measured as part of metabolic panel in milligrams per deciliter
Total Bilirubin | 2 weeks of assigned intervention
  Total bilirubin measured as part of metabolic panel in milligrams per deciliter
Blood urea nitrogen | baseline
  Blood urea nitrogen measured as part of metabolic panel in milligrams per deciliter
Blood urea nitrogen | 2 weeks of assigned intervention
  Blood urea nitrogen measured as part of metabolic panel in milligrams per deciliter
Calcium | baseline
  Calcium measured as part of metabolic panel in milligrams per deciliter
Calcium | 2 weeks of assigned intervention
  Calcium measured as part of metabolic panel in milligrams per deciliter
Carbon dioxide | baseline
  Carbon dioxide measured as part of metabolic panel in millimoles per liter
Carbon dioxide | 2 weeks of assigned intervention
  Carbon dioxide measured as part of metabolic panel in millimoles per liter
Chloride | baseline
  Chloride measured as part of metabolic panel in millimoles per liter.
Chloride | 2 weeks of assigned intervention
  Chloride measured as part of metabolic panel in millimoles per liter.
Creatinine | baseline
  Creatinine measured as part of metabolic panel in milligrams per deciliter
Creatinine | 2 weeks of assigned intervention
  Creatinine measured as part of metabolic panel in milligrams per deciliter
Estimated glomerular filtration rate | baseline
  Estimated glomerular filtration rate as part of metabolic panel in milliliters per minute per 1.73
Estimated glomerular filtration rate | 2 weeks of assigned intervention
  Estimated glomerular filtration rate as part of metabolic panel in milliliters per minute per 1.73
Blood Glucose | baseline
  Glucose measured as part of metabolic panel in milligrams per deciliter
Blood Glucose | 2 weeks of assigned intervention
  Glucose measured as part of metabolic panel in milligrams per deciliter
Potassium | baseline
  Potassium measured as part of metabolic panel in millimoles per liter.
Potassium | 2 weeks of assigned intervention
  Potassium measured as part of metabolic panel in millimoles per liter.
Sodium | baseline
  Sodium measured as part of metabolic panel in millimoles per liter.
Sodium | 2 weeks of assigned intervention
  Sodium measured as part of metabolic panel in millimoles per liter.
Total Globulin | baseline
  Total Globulin measured as part of metabolic panel in grams per deciliter
Total Globulin | 2 weeks of assigned intervention
  Total Globulin measured as part of metabolic panel in grams per deciliter
Total Protein | baseline
  Total Protein measured as part of metabolic panel in grams per deciliter
Total Protein | 2 weeks of assigned intervention
  Total Protein measured as part of metabolic panel in grams per deciliter
Albumin/globulin ratio | baseline
  Albumin/globulin ratio measured as part of metabolic panel
Albumin/globulin ratio | 2 weeks of assigned intervention
  Albumin/globulin ratio measured as part of metabolic panel
Blood urea nitrogen/creatinine ratio | baseline
  Blood urea nitrogen/creatinine ratio measured as part of metabolic panel
Blood urea nitrogen/creatinine ratio | 2 weeks of assigned intervention
  Blood urea nitrogen/creatinine ratio measured as part of metabolic panel
Hematocrit | baseline
  Hematocrit as part of a complete blood count panel measured as percentage
Hematocrit | 2 weeks of assigned intervention
  Hematocrit as part of a complete blood count panel measured as percentage
Hemoglobin | baseline
  Hemoglobin as part of a complete blood count panel measured in grams per deciliter
Hemoglobin | 2 weeks of assigned intervention
  Hemoglobin as part of a complete blood count panel measured in grams per deciliter
Mean corpuscular volume | baseline
  Mean corpuscular volume as part of a complete blood count panel measured in femtoliters
Mean corpuscular volume | 2 weeks of assigned intervention
  Mean corpuscular volume as part of a complete blood count panel measured in femtoliters
Mean corpuscular hemoglobin | baseline
  Mean corpuscular hemoglobin as part of a complete blood count panel measured in picograms
Mean corpuscular hemoglobin | 2 weeks of assigned intervention
  Mean corpuscular hemoglobin as part of a complete blood count panel measured in picograms
Mean corpuscular hemoglobin concentration | baseline
  Mean corpuscular hemoglobin concentration as part of a complete blood count panel measured in grams per deciliter
Mean corpuscular hemoglobin concentration | 2 weeks of assigned intervention
  Mean corpuscular hemoglobin concentration as part of a complete blood count panel measured in grams per deciliter
Red cell distribution width | baseline
  Red cell distribution width as part of a complete blood count panel measured as a percentage
Red cell distribution width | 2 weeks of assigned intervention
  Red cell distribution width as part of a complete blood count panel measured as a percentage
Platelets | baseline
  Platelets as part of a complete blood count panel measured as a count per 1000 per microliter
Platelets | 2 weeks of assigned intervention
  Platelets as part of a complete blood count panel measured as a count per 1000 per microliter
Specific gravity | baseline
  Specific gravity as measured as part of urinalysis (no units)
Specific gravity | 2 weeks of assigned intervention
  Specific gravity as measured as part of urinalysis (no units)
pH | baseline
  pH as measured as part of urinalysis (no units)
pH | 2 weeks of assigned intervention
  pH as measured as part of urinalysis (no units)
Urine color | baseline
  Urine color as reported as part of urinalysis (no units)
Urine color | 2 weeks of assigned intervention
  Urine color as reported as part of urinalysis (no units)
Urine Appearance | baseline
  Urine Appearance as reported as part of urinalysis (no units)
Urine Appearance | 2 weeks of assigned intervention
  Urine Appearance as reported as part of urinalysis (no units)
White Blood Cell esterase | baseline
  White blood cell esterase as measured as part of urinalysis, if present
White blood cell esterase | 2 weeks of assigned intervention
  White blood cell esterase as measured as part of urinalysis, if present
Protein | baseline
  Protein as measured as part of urinalysis, if present
Protein | 2 weeks of assigned intervention
  Protein as measured as part of urinalysis, if present
Glucose | baseline
  Glucose as measured as part of urinalysis, if present
Glucose | 2 weeks of assigned intervention
  Glucose as measured as part of urinalysis, if present
Ketones | baseline
  Ketones as measured as part of urinalysis, if present
Ketones | 2 weeks of assigned intervention
  Ketones as measured as part of urinalysis, if present
Occult blood | baseline
  Occult blood as measured as part of urinalysis, if present
Occult blood | 2 weeks of assigned intervention
  Occult blood as measured as part of urinalysis, if present
Bilirubin | baseline
  Bilirubin as measured as part of urinalysis, if present
Bilirubin | 2 weeks of assigned intervention
  Bilirubin as measured as part of urinalysis, if present
Urobilinogen | baseline
  Urobilinogen as measured as part of urinalysis in milligrams per deciliter
Urobilinogen | 2 weeks of assigned intervention
  Urobilinogen as measured as part of urinalysis in milligrams per deciliter
Microscopic examination | baseline
  Microscopic examination as reported as part of urinalysis, if indicated
Microscopic examination | 2 weeks of assigned intervention
  Microscopic examination as reported as part of urinalysis, if indicated
Total Cholesterol | baseline
  Total Cholesterol as reported as part of lipid panel in milligrams per deciliter
Total Cholesterol | 2 weeks of assigned intervention
  Total Cholesterol as reported as part of lipid panel in milligrams per deciliter
Triglycerides | baseline
  Triglycerides as reported as part of lipid panel in milligrams per deciliter
Triglycerides | 2 weeks of assigned intervention
  Triglycerides as reported as part of lipid panel in milligrams per deciliter
High-Density Lipoprotein Cholesterol | baseline
  High-Density Lipoprotein Cholesterol as reported as part of lipid panel in milligrams per deciliter
High-Density Lipoprotein Cholesterol | 2 weeks of assigned intervention
  High-Density Lipoprotein Cholesterol as reported as part of lipid panel in milligrams per deciliter
Very Low-Density Lipoprotein Cholesterol | baseline
  Very Low-Density Lipoprotein Cholesterol as reported as part of lipid panel in milligrams per deciliter
Very Low-Density Lipoprotein Cholesterol | 2 weeks of assigned intervention
  Very Low-Density Lipoprotein Cholesterol as reported as part of lipid panel in milligrams per deciliter
Low-Density Lipoprotein Cholesterol | baseline
  Low-Density Lipoprotein Cholesterol as reported as part of lipid panel in milligrams per deciliter
Low-Density Lipoprotein Cholesterol | 2 weeks of assigned intervention
  Low-Density Lipoprotein Cholesterol as reported as part of lipid panel in milligrams per deciliter
Mood questionnaire | baseline
  Visual analog scale used to assess mood (attentive, tired, alert, groggy, focused, sluggish, energetic, lethargic, fatigued, mental clarity, motivation, happiness, and feeling from 0 (None) to 10 (Extreme) as well as "Flushed out" from 0 (not at all) to 10 (completely empty)
Mood questionnaire | 2 weeks of assigned intervention
  Visual analog scale used to assess mood (attentive, tired, alert, groggy, focused, sluggish, energetic, lethargic, fatigued, mental clarity, motivation, happiness, and feeling from 0 (None) to 10 (Extreme) as well as "Flushed out" from 0 (not at all) to 10 (completely empty)
36-item short form survey | baseline
  36-item questionnaire that measures health-related quality of life with responses used to calculate scores on a scale of 0-100, where higher scores indicate better health.
36-item short form survey | 2 weeks of assigned intervention
  36-item questionnaire that measures health-related quality of life with responses used to calculate scores on a scale of 0-100, where higher scores indicate better health.
Tolerability Questionnaire | baseline
  18 item questionnaire covering upper abdominal, lower abdominal, and other symptoms using a 0-9 scale (0-no problem at all to 9-the worst it has ever been)
Tolerability Questionnaire | 1 day of assigned treatment
  18 item questionnaire covering upper abdominal, lower abdominal, and other symptoms using a 0-9 scale (0-no problem at all to 9-the worst it has ever been)
Tolerability Questionnaire | 3 days of assigned treatment
  18 item questionnaire covering upper abdominal, lower abdominal, and other symptoms using a 0-9 scale (0-no problem at all to 9-the worst it has ever been)
Tolerability Questionnaire | 1 week of assigned treatment
  18 item questionnaire covering upper abdominal, lower abdominal, and other symptoms using a 0-9 scale (0-no problem at all to 9-the worst it has ever been)
Tolerability Questionnaire | 2 weeks of assigned treatment
  18 item questionnaire covering upper abdominal, lower abdominal, and other symptoms using a 0-9 scale (0-no problem at all to 9-the worst it has ever been)
Bristol Chart | 3 days before baseline
  Self-reported number and consistency of daily bowel movements
Bristol Chart | 2 days before baseline
  Self-reported number and consistency of daily bowel movements
Bristol Chart | 1 day before baseline
  Self-reported number and consistency of daily bowel movements
Bristol Chart | 1 day of assigned treatment
  Self-reported number and consistency of daily bowel movements
Bristol Chart | 2 days on assigned treatment
  Self-reported number and consistency of daily bowel movements
Bristol Chart | 3 days of assigned treatment
  Self-reported number and consistency of daily bowel movements
Bristol Chart | 7 days of assigned treatment
  Self-reported number and consistency of daily bowel movements
Bristol Chart | 14 days of assigned treatment
  Self-reported number and consistency of daily bowel movements
Weight | baseline
  Body weight measured in kg
Weight | 2 weeks of assigned treatment
  Body weight measured in kg
Skin age | baseline
  a quantitative skin age based on skin parameters will be determined by the 3D P Plus system
Skin age | 2 weeks of assigned treatment
  a quantitative skin age based on skin parameters will be determined by the 3D P Plus system
Diastolic blood pressure | baseline
  Diastolic blood pressure will be measured using an automated blood pressure machine in units millimeters of mercury
Diastolic blood pressure | 2 weeks of assigned treatment
  Diastolic blood pressure will be measured using an automated blood pressure machine in units millimeters of mercury
Systolic blood pressure | baseline
  Systolic blood pressure will be measured using an automated blood pressure machine in units millimeters of mercury
Systolic blood pressure | 2 weeks of assigned treatment
  Systolic blood pressure will be measured using an automated blood pressure machine in units millimeters of mercury
Heart rate | baseline
  Heart rate will be measured using an automated blood pressure machine in units beats per minute
Heart Rate | 2 weeks of assigned treatment
  Hear rate will be measured using an automated blood pressure machine in units beats per minute

SECONDARY OUTCOMES:
Daily food diary | 3 days prior to baseline visit
  Daily food diary of all food and drink consumed that day
Daily food diary | 2 days prior to baseline visit
  Daily food diary of all food and drink consumed that day
Daily food diary | 1 day prior to baseline visit
  Daily food diary of all food and drink consumed that day
Daily food diary | 3 days prior to 2 week visit
  Daily food diary of all food and drink consumed that day
Daily food diary | 2 days prior to 2 week visit
  Daily food diary of all food and drink consumed that day
Daily food diary | 1 day prior to 2 week visit
  Daily food diary of all food and drink consumed that day

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States